CLINICAL TRIAL: NCT07058662
Title: A Phase 1/2, Open-label Clinical Study to Evaluate the Safety, Tolerability and Efficacy of BBM-D101 in the Treatment of Duchenne Muscular Dystrophy.
Brief Title: A Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of BBM-D101 in the Treatment of Duchenne Muscular Dystrophy.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Belief BioMed (Beijing) Co., Ltd (Industry)
Collaborators: Shanghai Mianyi Biopharmaceutical Co., Ltd. (Unknown); Shanghai Xinzhi BioMed Co., Ltd. (Industry); Belief BioMed Limited (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBM041-CLN1001
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: DMD
Keywords: DMD; gene therapy; Adeno-Associated Virus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm of BBM-D101 (Experimental): Single-dose treatment
  Interventions: Genetic: Single dose intravenous of BBM-D101

INTERVENTIONS:
Genetic: Single dose intravenous of BBM-D101 — BBM-D101 is a gene addition therapy based on engineered AAV delivery therapeutic protein gene cassette into muscle for treating DMD. Therapeutic protein could mediate the dystrophin-associated protein complex to prevent muscular dystrophy and to rescue the function of muscle.The administration is completed by a single intravenous infusion.

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and efficacy of BBM-D101 to treat participants with Duchenne Muscular Dystrophy.

DETAILED DESCRIPTION:
This is a single-arm, open-label study to evaluate the safety, tolerability, efficacy, pharmacokinetic, pharmacodynamic, and immune response of BBM-D101 within 52 weeks after a single intravenous infusion in DMD boys, as well as the long-term safety and efficacy of BBM-D101 for up to 5 years post infusion.

BBM-D101 is a gene addition therapy based on engineered AAV delivery therapeutic protein gene cassette into muscle for treating DMD. Therapeutic protein could mediate the dystrophin-associated protein complex to prevent muscular dystrophy and to rescue the function of muscle.

ELIGIBILITY:
Inclusion Criteria:

1. The Participants and/or his legal guardian must fully understand the purpose, nature, methods, and potential risks of the study, and sign a written informed consent form.
2. Ambulatory male subjects aged 4 years and above but under 9 years (4 years ≤ age < 9 years).
3. Any mutation in the DMD gene confirmed by genetic testing
4. Serum creatine kinase (CK) during the screening period meets the study requirements.
5. Receiving stable, standard-dose glucocorticoids before screening.
6. The subject's AAV capsid antibodies meet the clinical trial requirements.
7. Able to cooperate with motor function assessment, MRI, and muscle biopsy as required by the study.
8. Laboratory test results during the screening period and at baseline meet the standards.
9. The subject and/or his legal guardian must fully understand the study procedures, be willing to actively cooperate, commit to high compliance with the protocol, and ensure that the subject attends all scheduled visits.

Exclusion Criteria:

1. Positive for hepatitis B surface antigen (HBsAg), hepatitis B virus deoxyribonucleic acid (HBV-DNA) ≥ 1000 U/mL, hepatitis C virus ribonucleic acid (HCV-RNA) positive, human immunodeficiency virus (HIV) positive, or positive for Treponema pallidum antibodies.
2. Currently receiving antiviral therapy for hepatitis B, hepatitis C, HIV, etc.
3. The investigator deems the subject has severe behavioral or cognitive disorders that may hinder participation in this study.
4. Poorly controlled asthma, or Duchenne Muscular Dystrophy (DMD) leading to significant decline in lung function, or recurrent infectious pneumonia that the investigator considers may affect respiratory function.
5. Left ventricular ejection fraction (LVEF) < 50% or New York Heart Association (NYHA) cardiac function class ≥ III.
6. Severe or persistent arrhythmias (such as atrial fibrillation, frequent ventricular premature beats, ventricular bigeminy, ventricular trigeminy, severe bundle branch block, etc.), and congenital heart disease that is evaluated by the investigator as unsuitable for participation in this study.
7. Any changes in preventive/cardiomyopathy treatment (initiation of treatment, drug changes, dosing regimen changes, treatment interruption, termination, or restart) within 1 month before the infusion of the study drug.
8. History of liver diseases such as portal hypertension, splenomegaly, hepatic encephalopathy, liver fibrosis ≥ stage 3, or hepatic nodules/cysts found by ultrasound during screening, or elevated alpha-fetoprotein with clinical significance as determined by the investigator.
9. Severe infection (such as pneumonia, pyelonephritis, or meningitis) within 4 weeks before the treatment visit (enrollment may be postponed).
10. History of gene therapy or cell therapy (such as stem cell transplantation).
11. History of or current presence of autoimmune diseases, severe renal, gastrointestinal, neurological, or coagulation disorders, malignant tumors, or other diseases.
12. Other diseases that the investigator deems unsuitable for participation in this study.

Ages: 4 Years to 9 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) events | Within 12 weeks
  To evaluate the rate of incidence of DLT events determined by the Safety Data Review Committee (SRC) in DLT observation period after BBM-D101 infusion.
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Within 12 weeks
  To evaluate the safety of BBM-D101 by AEs and SAEs.

SECONDARY OUTCOMES:
Changes from baseline in BBM-D101 therapeutic protein level of muscle biopsy samples | Within 52 weeks
  To assess changes of therapatic protein from baseline in muscle after BBM-D101 Infusion.
Changes from baseline in serum Creatine Kinase (CK) level | Within 52 weeks
  To assess changes of serum CK after BBM-D101 Infusion.
Changes from baseline in the time to ascend time to rise (TTR) without assistance | Within 52 weeks
  To assess changes in TTR from baseline within 52 weeks after BBM-D101 infusion.
Changes from baseline in the time to ascend 10-meter walk/run test (10MWR) without assistance | Within 52 weeks
  To assess changes in 10MWR from baseline within 52 weeks after BBM-D101 infusion.
Changes from baseline in the time to ascend 4 steps (4-stair climb, 4-SC) without assistance. | Within 52 weeks
  To assess changes in 4-SC from baseline within 52 weeks after BBM-D101 infusion.
Changes from baseline in the North Star Ambulatory Assessment (NSAA). | Within 52 weeks
  To assess changes in NSAA from baseline within 52 weeks after BBM-D101 infusion; The NSAA is a scale that rates performance of various motor abilities in ambulant children with Duchenne Muscular Dystrophy and is used to monitor disease progression and treatment effects. The NSAA total score is defined as the sum of all 17items, ranging from 0 (worst) to 34 (best).
Changes from baseline in the TTR， 10MWR , 4-SC，NSAA. | Within 5 years
  Evaluate the changes from baseline in TTR, 10MWR, 4-SC and NSAA in Participants after Infusion of BBM-D101.
Incidence of AEs and SAEs. | Within 5 years
  To assess the long-term safety of BBM-D101 by AEs and SAEs.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Dai, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No